CLINICAL TRIAL: NCT01234623
Title: Pilot Phase. Cord Blood Serum in the Treatment of Ocular Surface Diseases
Brief Title: Cord Blood Serum in the Treatment of Ocular Surface Diseases
Status: Completed | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Emilio C Campos, Head. Ophthalmology Unit
Other Study IDs: EudraCT: 2008-005757-38
Record Dates: First submitted 2010-10-12; First posted 2010-11-04 (Estimated); Last update posted 2011-05-26 (Estimated); Status verified 2011-04

CONDITIONS: Graft vs Host Disease; Sjogren's Disease
Keywords: Umbilical cord serum, eyedrops, GVHD, SS-I, corneal healing
MeSH Terms: conditions — Graft vs Host Disease; Sjogren's Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- UCB eyedrops, single arm: One-centre pilot study, open, non randomized.
  Interventions: Other: UCS eyedrops

INTERVENTIONS:
Other: UCS eyedrops — 1 ml UCS eyedrops/day topically applied 8 times/day 1 drop/eye for 28 days
  Other Names: no brand names, serial or code numbers

SUMMARY:
Human autologous serum (AS) eye drops have been successfully used in the treatment of severe ocular surface disorders and the enhancement of corneal wound healing, due to their growth factor (GF) content. Umbilical cord serum (UCS) contains even higher GF concentrations and the objective of the study was to prove whether UCS eye drops

1. are effective in the healing of corneal epithelial defects.
2. ameliorate the painful subjective symptoms

DETAILED DESCRIPTION:
The regular collection and banking of cord blood remaining in the placenta after baby's delivery started in the early 1990s and was prompted by the observation that cord blood shows an immunological immaturity which allows to avoid any matching between donor-mother source and patient-recipient, it contains a number of haemopoietic progenitor and stem cells and is therefore potentially and safely useful in the field of regenerative medicine.

Cord blood collection occurs after the umbilical cord has been cut and is extracted from the fetal end of the cord. After collection, the cord blood unit bag is delivered to the lab, processed and then cryopreserved.

The main current clinical use of cord blood is allogeneic transplantation in patients suffering from severe blood diseases but physicians and researchers are making significant progresses evaluating the safety and efficacy of umbilical cord blood stem cells for therapeutic uses far beyond their uses for blood disorders.

Umbilical cord serum (UCS) contains many growth factors and especially EGF and TGF-beta1 concentrations are two-three times higher than in peripheral blood serum and much higher than in tears and is sufficient to prevent squamous metaplasia. In addition, UCS contains anti-inflammatory cytokines with protective effect.

Current therapy for SS-I and GVHD related dry eye depends upon clinical severity of the disease. From mild to progressively severe involvement of corneal epithelial damage , tear substitutes, FANS, steroids, Cyclosporin A, contact lens shields can be topically applied alone or in combination. Autologous serum eyedrops can be an option in severe cases as well, since it supplies epithelial growth factors to the healing process of epithelium.

The use of autologous serum eyedrops, however, is a controversial issues in diseases where inflammatory cytokines are present in peripheral blood, such as GVHD.

The use of cord blood serum based tear substitutes has been recently proposed in the literature for the treatment of ocular surface diseases and neurotrophic keratitis, because it contains growth factors, neurotrophic factors and essential components of tears. Moreover, serum from cord blood is readily available from cord blood banks as quality controlled product and is therefore theoretically attractive for topical use in ophthalmology.

The use of cord blood serum eyedrops as a biological preparation can display in itself efficacy features higher than the other drugs in terms of healing and anti-inflammatory properties in absence of any chemical compound.

In Italy biological products for topical use in ophthalmology to treat corneal epithelial severe defects are not available. The originality of the present study is based on the optimization and standardization of biological eyedrops prepared from cord blood serum. The efficacy and safety of the product for topical use in ocular surface diseases will be evaluated .

For the purpose, the following methods will be applied at baseline and endpoint (28 days of treatment with UCS eyedrops):

1. Patients' subjective symptoms evaluation by a validated questionnaire for dry eye (OSDI)
2. Slit Lamp examination and evaluation of Tear Film Break Up Time, corneal fluorescein staining score, conjunctival lissamine green staining score, staining will be recorded with digital photos to estimate the healing area in the follow up
3. Schirmer I test to evaluate tear production
4. Corneal sensitivity test (measured with a Cochet-Bonnet esthesiometer)
5. Tear osmolarity, (TearLab, TearLab S.Diego) an indicator of the ability of the patient to compensate
6. Tear Clearance Rate, a global indicator of tear production and tear evaporation
7. Tear Proteomic to evaluate tear protein profile
8. Corneal and Conjunctival inflammatory marker evaluation on cells collected by imprint and scraping cytology

Data will be statistically evaluated after 28 days treatment and matched vs baseline by using the descriptive statistics for paired data. Statistic outcomes will be analyzed with caution due to the non-randomized study design.

ELIGIBILITY:
Inclusion Criteria:

* to suffer from GVHD after bone marrow transplantation or SS-I
* presence of permanent or transient corneal epithelial defects scored > 2 , according to DEWS severity classification
* to be in a general healthy condition
* signature of study consent for participation and personal data treatment.

Exclusion Criteria:

* to suffer from glaucoma and being under treatment with antiglaucomatous drugs
* to have received refractive surgery over the past year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult outpatients suffering from ocular surface discomfort and recurrent or permanent corneal epithelial defects
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2010-02; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Corneal epithelial damage evaluated by fluorescein staining (micron meter squares) with digital photos | 28 days treatment
  Digital photographs taken at the slit lamp will be evaluated by means of an Image Analyzer softare, to determine the area of corneal epithelial damage involved at a given stand point. Reduction of damaged area will be estimated in micron meter squares

SECONDARY OUTCOMES:
Reduction the patients' painful subjective symptoms | 28 days treatment
  Subjective symptoms will be evaluated by means of a validated Questionnaire (OSDI, Ocular Surface Disease Index) at the given stand points
Reduction the patients' painful subjective symptoms | 15 days treatment
  Subjective symptoms will be evaluated by means of a validated Questionnaire (OSDI, Ocular Surface Disease Index) at the given stand points

CONTACTS AND LOCATIONS:
Overall Officials: Emilio C Campos, MD, Study Director — Head of Ophthalmology Unit, Dept.of Specialistic Surgery and Anesthesiological Sciences, University of Bologna, Policlinico S. Orsola-Malpighi, Pad 1 Palagi, Via Palagi 9 -40138 Bologna Italy
Locations (1):
- Ophthalmology Unit, Dept.of Specialistic Surgery and Anesthesiological Sciences, Bologna, Bologna, Italy

REFERENCES:
- [Background] Buzzi M, Versura P, Vaselli C, Coslovi C, Terzi A, Bontadini A, Campos EC. Fattori di crescita epiteliali nel sangue cordonale. SIES 2008, Bari 24-26 settembre 2008, abstract
- [Result] P. Versura, V. Profazio, L. Foroni, M. Buzzi, A. Stancari, EC Campos. Cord blood serum eye drops in the treatment of ocular surface diseases in GVHD patients. A pilot study. 6th International Conference on the Tear Film & Ocular Surface: Basic Science and Clinical Relevance, Florence , September 22-25, 2010 Abstract
- [Derived] Versura P, Profazio V, Buzzi M, Stancari A, Arpinati M, Malavolta N, Campos EC. Efficacy of standardized and quality-controlled cord blood serum eye drop therapy in the healing of severe corneal epithelial damage in dry eye. Cornea. 2013 Apr;32(4):412-8. doi: 10.1097/ICO.0b013e3182580762. PMID 22955120